CLINICAL TRIAL: NCT00921479
Title: Postoperative Course and Quality of Life Following Surgical Removal of the Mandibular 3. Molar
Brief Title: Postoperative Course Following Wisdom Tooth Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ullevaal University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Lasse Ansgar Skoglund, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Other Study IDs: OE-001
Record Dates: First submitted 2009-06-09; First posted 2009-06-16 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Pain, Postoperative
Keywords: third molar; quality of life; postoperative swelling; postoperative pain; Surgical Procedures, Operative; Postoperative Period
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Females: Norwegian females Caucasian origin, between the age of 18 and 45, who are candidates for surgical removal of one mandibular 3. molar.
- Males: Norwegian males of Caucasian origin, between the age of 18 and 45, who are candidates for surgical removal of one mandibular 3. molar

SUMMARY:
The purpose of this study is to determine how quality of life changes after surgical removal of wisdom teeth

DETAILED DESCRIPTION:
A significant percentage of patients are subjected to surgical removal of 3. molars every year. The surgical mucosal and osseous procedure may lead to postoperative discomfort including pain, for the patient. Information with respect to how patients regard the impact of this surgical treatment on oral health including pain and swelling is of great interest. More precise information about the postoperative course following this surgery will be beneficial in improving clinical treatment procedures with respect to alleviating the patients' postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex of Caucasian origin, between the age of 18 and 45, who are candidates for surgical removal of one mandibular 3. molar

Exclusion Criteria:

* Chronic drug treatment (except birth control medication) with analgesics, anti-inflammatory treatment (both steroidal (SAIDs) and non-steroidal anti-inflammatory drugs (NSAIDs)) apart from standard postoperative analgesic treatment administered by the operator.
* The necessity for anti-microbial drugs.
* Pregnant or lactating women.
* Patients with diabetes.
* Patients who due to age or communication skills are considered unable to complete patient forms.
* Professional evaluation suggests an alteration of the planned surgical area or treatment form.
* Surgery exceeding 45 minutes, from time of first incision to completed suturing.
* Known or assumed intolerance or hypersensibility to ibuprofen (standard postoperative analgesic treatment).
* Known or assumed intolerance or hypersensibility to the standard local anaesthetic Xylocain-adrenalin (lidocaine-adrenalin).
* Consumption of alcohol in the period from 2 days before or until the end of the primary observation period (postoperative days 0-7.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Norwegian outpatients patients of Caucasian origin operated in a primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-06; Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral Health Impact Profile (OHIP-14) | 7 days
  Measure functional status of the oral cavity

SECONDARY OUTCOMES:
Pain Intensity (0-10 Numerical Rating Scale) | 7 days
  Subjective measure pain intensity
Norwegian McGill Pain Questionnaire (NMPQ) | 7 days
  Measure quantitative and qualitative pain characteristics
Norwegian Translated Short-Form McGill Pain Questionnaire (NTSF-MPQ) | 7 days
  Measure qualitative and quantitative pain characetristics
Subjective Swelling Assessment (0-10 Numerical rating Scale) | 7 Days
  Subjective assessment of postoperative swelling
Corahs Dental Anxiety Scale (CDAS) | 1 day
  Assessment of preoperative anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Lasse A Skoglund, DDS, DSci, Principal Investigator — Section of Dental Pharmacology and Pharmacotherapy, Faculty of Dentistry, University of Oslo
Locations (2):
- Norway (2):
  - Department of Oral and Maxillofacial Surgery, Ullevaal University Hospital, Oslo
  - Department of Oral and Maxillofacial Surgery, OUS, Oslo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coll AM, Ameen JR, Mead D. Postoperative pain assessment tools in day surgery: literature review. J Adv Nurs. 2004 Apr;46(2):124-33. doi: 10.1111/j.1365-2648.2003.02972.x. PMID 15056325
- [Background] Corah NL. Dental anxiety. Assessment, reduction and increasing patient satisfaction. Dent Clin North Am. 1988 Oct;32(4):779-90. PMID 3053270
- [Background] Kim HS, Schwartz-Barcott D, Holter IM, Lorensen M. Developing a translation of the McGill pain questionnaire for cross-cultural comparison: an example from Norway. J Adv Nurs. 1995 Mar;21(3):421-6. doi: 10.1111/j.1365-2648.1995.tb02722.x. PMID 7745193
- [Background] Melzack R. The short-form McGill Pain Questionnaire. Pain. 1987 Aug;30(2):191-197. doi: 10.1016/0304-3959(87)91074-8. PMID 3670870
- [Background] Melzack R. The McGill Pain Questionnaire: major properties and scoring methods. Pain. 1975 Sep;1(3):277-299. doi: 10.1016/0304-3959(75)90044-5. PMID 1235985
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Slade GD. Assessing change in quality of life using the Oral Health Impact Profile. Community Dent Oral Epidemiol. 1998 Feb;26(1):52-61. doi: 10.1111/j.1600-0528.1998.tb02084.x. PMID 9511843